CLINICAL TRIAL: NCT03384875
Title: CytoSorb® Reduction of FREee Hemoglobin/Acute Kidney Injury (AKI) During Cardiac Surgery (REFRESH II Trial)
Brief Title: CytoSorb® Reduction of FREee Hemoglobin/Acute Kidney Injury (AKI) During Cardiac Surgery
Acronym: REFRESH II-AKI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision for business reasons
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-001
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2022-08

CONDITIONS: Elective Cardiac Surgery
Keywords: CytoSorb device; Plasma free hemoglobin; inflammation; extracorporeal cardiopulmonary bypass; cardiopulmonary bypass; Acute Kidney Injury
MeSH Terms: conditions — Inflammation; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CytoSorb Device (Experimental): Standard of care plus treatment with CytoSorb device installed on the Cardiopulmonary bypass (CPB) machine
  Interventions: Device: CytoSorb
- Control (Placebo Comparator): Standard of care
  Interventions: Device: CytoSorb

INTERVENTIONS:
Device: CytoSorb — To evaluate the safety and performance of the CytoSorb® device to decrease the incidence or severity of acute kidney injury (AKI)
  Other Names: CytoSorb device used during cardiopulmonary bypass (CPB)

SUMMARY:
Prospective, multi-center, randomized, blinded, pivotal clinical study. Subjects will be randomized in a 1:1 ratio to either standard of care (SOC) alone or standard of care plus treatment with the CytoSorb® device.

DETAILED DESCRIPTION:
To evaluate the safety and performance of the CytoSorb® device to decrease the incidence or severity of acute kidney injury (AKI) as defined by Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guideline definition of acute kidney injury when used intraoperatively with cardiopulmonary bypass (CPB) in subjects undergoing cardiac surgery. The objective of using CytoSorb® treatment in this setting is to provide clinically meaningful improvements in renal function by mitigation of intraoperative injury by removal of nephrotoxic agents such as pfHb and complement. Up to 420 subjects will be enrolled and randomized at a 1:1 ratio at up to 40 investigational sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for non-emergent cardiac surgery requiring CPB for i) heart valve replacement with any other procedure, without hypothermic circulatory arrest (HCA), or ii) aortic reconstruction with or without another procedure, with HCA

Exclusion Criteria:

* Isolated Coronary Artery Bypass Graft
* Pregnant women
* Life expectancy of < 14 days
* End stage organ disease
* Active infection
* Correction of a congenital heart defect
* Contraindication to anticoagulation with heparin
* Minimally invasive surgery implantation (TAVI) or transcatheter aortic valve replacement (TAVR)
* Declined informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gleason, MD, Principal Investigator — not applicable- Unaffiliated with CytoSorbents
Locations (20):
- United States (20):
  - Yale School of Medicine, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Louisville, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Valley Hospital, Ridgewood, New Jersey
  - Columbia University Medical Center, New York, New York
  - Northwell Health: Lennox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - The Christ Hospital Linder Research Center, Cincinnati, Ohio
  - Ohio State university, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 Subjects exited study post consent, but pre-procedure: 21 of these were screen failures (20 did not meet eligibility criteria, 1 was reported as Screen failure for reasons other than not meeting the eligibility criteria).
  4 were withdrawn due to investigator decision. 2 withdrew consent. 7 exited due to "other reasons."
Groups:
- Roll in: SOC + CytoSorb Device: Unblinded Standard of care plus treatment with CytoSorb device installed on the Cardiopulmonary bypass (CPB) machine
  CytoSorb: To evaluate the safety of the CytoSorb® device to decrease the incidence or severity of acute kidney injury (AKI)
Period: Overall Study
Arm/Group | CytoSorb Device | Control | Roll in: SOC + CytoSorb Device
Started | 56 (56 patients were randomized to Treatment Arm (SOC + CytoSorb Device); evaluated for all end points vs Control arm.) | 60 | 36 (36 patients were "Roll in"- First 2 subjects @ each site, automatically assigned to SOC + CytoSorb device as learning, evaluated for Safety, but not for efficacy.)
Completed | 54 | 59 | 36
Not Completed | 2 | 1 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Reason not provided | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Roll In: CytoSorb Device: Unblinded: Standard of care plus treatment with CytoSorb device installed on the Cardiopulmonary bypass (CPB) machine
  CytoSorb: To evaluate the safety and performance of the CytoSorb® device to decrease the incidence or severity of acute kidney injury (AKI)
- Total: Total of all reporting groups
Arm/Group | CytoSorb Device | Control | Roll In: CytoSorb Device | Total
Number analyzed (Participants) | 56 | 60 | 36 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.98 (11.87) | 64.10 (11.88) | 66.14 (11.84) | 65.64 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 9 | 45
  Male | 38 | 42 | 27 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 53 | 57 | 32 | 142
  Unknown or Not Reported | 2 | 1 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 3 | 10
  White | 51 | 56 | 31 | 138
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 56 | 60 | 36 | 152
Smoking History [Number; unit: participants]
  Current Smoker | 10 | 2 | 3 | 15
  Former Smoker | 19 | 28 | 16 | 63
  Never Smoked | 27 | 30 | 17 | 74

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Acute Kidney Injury (AKI) in the First 48 Hours After Cardiopulmonary Pulmonary Bypass (CPB)
Description: Incidence and severity of AKI in the first 48 hours after CPB, evaluated based on creatinine levels at CPB, 24 & 48h after CPB and urine output up to 48h.
Time Frame: From start of CPB through 48 hours after CPB
Measure: Count of Participants; unit: Participants
Arm/Group | CytoSorb Device | Control | Roll In: CytoSorb Device
Number analyzed (Participants) | 56 | 60 | 36
Participants
  AKI Stage 0 | 9 | 12 | 7
  AKI Stage 1 (Mild) | 7 | 5 | 2
  AKI Stage 2 (moderate) | 31 | 28 | 21
  AKI Stage 3 (Severe) | 9 | 15 | 6
Statistical Analysis 1: Comparison: CytoSorb Device vs Control; Test type: Superiority; p = 0.517, Chi-squared; Risk Difference (RD) = 0

2. Secondary Outcome: Summary of Health Resource Utilization: ICU Duration (Hours)
Description: Analysis of health resource utilization included parameters such as length of stay in ICU and hospital and need for supportive care measures such as vasopressors, and mechanical ventilation.
Time Frame: From start of CPB through discharge, average of 8.9 days.
Population: safety population analysis. Not all patients' data complete.
Measure: Median (Standard Deviation); unit: hours
Arm/Group | CytoSorb Device | Control | Roll in: SOC + CytoSorb Device
Number analyzed (Participants) | 56 | 60 | 36
hours | 70.63 (85.55) | 53.57 (67.60) | 66.83 (132.87)

3. Secondary Outcome: Summary of Health Resource Utilization: Post-Op Hospital Stay: Date of Discharge - Date of ICU Admission
Description: as for outcome 2
Time Frame: From start of CPB through discharge, average of 8.9 days.
Population: safety population analysis. Not all patients' data complete.
Measure: Median (Standard Deviation); unit: days
Arm/Group | CytoSorb Device | Control | Roll in: SOC + CytoSorb Device
Number analyzed (Participants) | 54 | 59 | 35
days | 8 (3.9) | 7 (4.7) | 7 (5.2)

4. Secondary Outcome: Summary of Health Resource Utilization: Number of Patients on Vasopressor Medication
Description: as for outcome 2
Time Frame: From start of CPB through discharge, average of 8.9 days.
Population: safety population analysis. Not all patients' data complete.
Measure: Count of Participants; unit: Participants
Arm/Group | CytoSorb Device | Control | Roll in: SOC + CytoSorb Device
Number analyzed (Participants) | 56 | 60 | 36
Participants | 44 | 48 | 32

5. Secondary Outcome: Summary of Health Resource Utilization: Duration of Continuous Intra-op to Post-op Ventilator/ Mechanical Support Use
Description: as for outcome 2
Time Frame: From start of CPB through discharge, average of 8.9 days.
Population: safety population analysis. Not all patients' data complete.
Measure: Median (Standard Deviation); unit: hours
Arm/Group | CytoSorb Device | Control | Roll in: SOC + CytoSorb Device
Number analyzed (Participants) | 56 | 60 | 36
hours | 12.83 (19.12) | 11.62 (60.38) | 13.30 (77.73)

6. Secondary Outcome: Initiation of Renal Replacement Therapy
Description: Initiation of Renal Replacement Therapy up to 48 Hours post CPB
Time Frame: Up to 48 hours after CPB
Measure: Count of Participants; unit: Participants
Arm/Group | CytoSorb Device | Control | Roll In: CytoSorb Device
Number analyzed (Participants) | 56 | 60 | 36
Participants | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of Consent to 30 days post-procedure +/- 5 days.
Description: Throughout the study, the Investigator or designee determined adverse event (AE) occurrences through assessment & regular laboratory testing.
Arm/Group | CytoSorb Device | Control | Roll in: SOC + CytoSorb Device
All-Cause Mortality (participants affected / at risk) | 1/56 | 1/60 | 0/36
Serious Adverse Events (participants affected / at risk) | 28/56 | 21/60 | 14/36
Other Adverse Events (participants affected / at risk) | 35/56 | 44/60 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CytoSorb Device (N=56) | Control (N=60) | Roll in: SOC + CytoSorb Device (N=36)
Atrial fibrillation (Cardiac disorders) | 6 (7) | 7 (7) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 5 (5) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 7 (7) | 3 (3) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CytoSorb Device (N=56) | Control (N=60) | Roll in: SOC + CytoSorb Device (N=36)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 9 (9) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 7 (7) | 10 (10)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 10 (10) | 6 (6) | 9 (9)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Acute Kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (3)
Acute respiratory failure (Renal and urinary disorders) | 4 (4) | 6 (6) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03384875/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03384875/SAP_001.pdf